CLINICAL TRIAL: NCT00388999
Title: Multi-Center,Open-Label,Randomized,Phase 1B Study Evaluating Safety & Tolerability of Intravenous rhMBL in Pts With Multiple Myeloma Receiving Melphalan-Based High-Dose Chemotherapy Followed by Autologous Hematopoietic Stem Cell Transplant
Brief Title: Intravenous rhMBL in Patients With Multiple Myeloma Receiving Chemotherapy Followed by Stem Cell Transplant
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Enzon Pharmaceuticals, Inc. (Industry)
Responsible Party: Nazish Huq, Clinical Project Manager, Enzon Pharmaceuticals, Inc
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EZN-2232-01
Record Dates: First submitted 2006-10-13; First posted 2006-10-17 (Estimated); Last update posted 2011-12-05 (Estimated); Status verified 2011-12

CONDITIONS: Multiple Myeloma
Keywords: Multiple Myeloma; Stem Cell Transplant; rhMBL
MeSH Terms: conditions — Multiple Myeloma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- 0 mg/kg (Other)
  Interventions: Drug: Intravenous Recombinant Human Mannose-Binding Lectin (rhMBL)
- 0.5 mg/kg (Other)
  Interventions: Drug: Intravenous Recombinant Human Mannose-Binding Lectin (rhMBL)
- 1.0 mg/kg (Other)
  Interventions: Drug: Intravenous Recombinant Human Mannose-Binding Lectin (rhMBL)

INTERVENTIONS:
Drug: Intravenous Recombinant Human Mannose-Binding Lectin (rhMBL) — Intravenous (i.v.) administration for 4 weeks. Patients will be randomized to one of three cohorts: 0 mg/kg; 0.5 mg/kg, or 1.0 mg.kg
  Arms: 0 mg/kg
Drug: Intravenous Recombinant Human Mannose-Binding Lectin (rhMBL) — Intravenous (i.v.) administration for 4 weeks. Patients will be randomized to one of three cohorts: 0 mg/kg; 0.5 mg/kg, or 1.0 mg.kg
  Arms: 0.5 mg/kg
Drug: Intravenous Recombinant Human Mannose-Binding Lectin (rhMBL) — Intravenous (i.v.) administration for 4 weeks. Patients will be randomized to one of three cohorts: 0 mg/kg; 0.5 mg/kg, or 1.0 mg.kg
  Arms: 1.0 mg/kg

SUMMARY:
MBL deficient patients enrolled in this protocol are scheduled to be treated with melphalan-based high-dose chemotherapy followed by autologous hematopoietic stem cell transplant (HSCT) for their multiple myeloma. Patients are randomized to 0.5 mg/kg, 1.0 mg/kg, or no rhMBL.

DETAILED DESCRIPTION:
MBL deficient patients will be randomized in a ratio of 2:2:1 to receive up to 4 weekly i.v. infusions of rhMBL at a dose of 0.5 mg/kg or 1.0 mg/kg, or standard anti-infectious prophylactic therapy alone. A total of 20 patients will be treated in each of the rhMBL arms, and 10 patients will receive best standard supportive prophylactic therapy but not rhMBL. All patients are to receive anti-infectious prophylactic supportive therapy as per institutional standards.

ELIGIBILITY:
Major Inclusion Criteria: Patients must meet all of the following criteria to be eligible for enrollment into the study:

* Capable of understanding the protocol requirements and risks and providing written informed consent.
* Histologically or cytologically confirmed diagnosis of multiple myeloma.
* Mannose-binding lectin level <300 ng/mL.
* Age ≥18 years old.
* Score of 0 to 2 on the Zubrod performance status scale.
* Patient is scheduled to receive melphalan-based high-dose chemotherapy and autologous HSCT for the treatment of multiple myeloma.

Exclusion Criteria:

* Concurrent serious medical illness that could potentially interfere with protocol compliance.
* Concurrent or previous malignancy associated with a poor prognosis.
* Known chronic infectious disease, such as acquired immunodeficiency syndrome (AIDS) or hepatitis (for hepatitis and human immunodeficiency virus [HIV] will not be performed).
* Positive screening pregnancy test or is breast-feeding.
* Female or male patient of reproductive capacity unwilling to use methods appropriate to prevent pregnancy during the course of this protocol.
* Known or clinically suspected active brain metastases.
* Current participation in another clinical study with an investigational agent and/or use of an investigational drug.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2006-09; Primary Completion 2009-02 (Actual); Study Completion 2009-05 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability of rhMBL | 2 months

SECONDARY OUTCOMES:
Pharmacokinetic (PK) of rhMBL | 2 months
Pharmacodynamics (PD) of rhMBL | 2 months
Immunogenicity of rhMBL, incidence of infectious complications | 2 months

CONTACTS AND LOCATIONS:
Overall Officials: Elias Anaissie, MD, Principal Investigator — University of Arkansas
Locations (1):
- University of Arkansas for Medical Sciences, Little Rock, Arkansas, United States